CLINICAL TRIAL: NCT04936581
Title: Patient Reported Outcomes Following Cancer of the Rectum
Acronym: PROCaRe
Status: Recruiting | Type: Observational
Sponsor: University Hospital Gregorio Marañón (Other)
Collaborators: University of Navarrra Hospital (Clinica Universitaria) (Other); Hospital de Leon (Other Government); Hospital del Rio Hortega (Other)
Responsible Party: Principal Investigator, Patricia Tejedor, Principal Investigator, University Hospital Gregorio Marañón
Other Study IDs: 205/15; NCT06290960 (obsolete NCT alias)
Record Dates: First submitted 2021-06-09; First posted 2021-06-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Sphincter Ani Incontinence; Rectal Cancer
Keywords: rectal cancer; taTME; laparoscopic TME; robotic TME; open TME; low anterior resection syndrome
MeSH Terms: conditions — Rectal Neoplasms; Low Anterior Resection Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Open Total Mesorectal Excision: Patients undergoing open low anterior resection
  Interventions: Procedure: Open Total Mesorectal Excision
- Laparoscopic Total Mesorectal Excision: Patients undergoing laparoscopic low anterior resection
  Interventions: Procedure: Laparoscopic Total Mesorectal Excision
- Robotic Total Mesorectal Excision: Patients undergoing robotic low anterior resection
  Interventions: Procedure: Robotic Total Mesorectal Excision
- Transanal Total Mesorectal Excision: Patients undergoing transanal Total Mesorectal Excision (taTME)
  Interventions: Procedure: Transanal Total Mesorectal Excision

INTERVENTIONS:
Procedure: Open Total Mesorectal Excision — Open approach for Total Mesorectal Excision
  Groups: Open Total Mesorectal Excision
Procedure: Laparoscopic Total Mesorectal Excision — Laparoscopic approach for Total Mesorectal Excision
  Groups: Laparoscopic Total Mesorectal Excision
Procedure: Robotic Total Mesorectal Excision — Robotic approach for Total Mesorectal Excision
  Groups: Robotic Total Mesorectal Excision
Procedure: Transanal Total Mesorectal Excision — Transanal approach for Total Mesorectal Excision
  Groups: Transanal Total Mesorectal Excision

SUMMARY:
The surgical management of rectal cancer includes a Total Mesorectal Excison (TME); depending on the height of the tumor, the problem of preservation of the anal sphincter arises, being able to perform a low anterior resection, an ultra-low anterior resection (RAUB) or an intersphincteric dissection. In some cases invading the sphincters or the puborectalis muscle, an abdominoperineal resection needs to be performed, being the gold standard in this particular situation so far.

TME can be performed by open, laparoscopic, robotic or transanal approaches, as long as the oncological principles for the resection are achieved. Unfortunately, up to 90% of these patients will present a change in bowel habit, ranging from an increased frequency of bowel movements to the degree of fecal incontinence or evacuation dysfunction. Of these patients, 25-50% will have a severe alteration in the quality of life. This wide spectrum of symptoms has been called "low anterior resection syndrome" (LARS). Other collateral damage is the change in sexual and urinary function, due to hypogastric plexus injury. There is a significant lack of multicenter prospective studies that provide evidence, and that reveal the functional results and quality of life of these techniques available to date for the management of rectal cancer.

The study is set up as a prospective multicentre observational study. Inclusion criteria are: 1) patients over 18 years old, 2) diagnosed with rectal cancer located below the peritoneal reflection, defined by preoperative MRI, 3) undergoing Open, laparoscopic, robotic or Transanal Total Mesorectal Excision (taTME) approaches, 4) with/without derivative stoma and 5) with/without neoadjuvant treatment. Exclusion criteria are: 1) Upper rectal cancer, located above the peritoneal reflection, 2) previous radical prostatectomy, 3) previous pelvic radiotherapy, 4) rectal resection without primary anastomosis, 5) intraoperative findings of peritoneal carcinomatosis, 6) stage IV disease, 7) multivisceral or en-bloc resection, which includes uterus, prostate, vagina or bladder, 8) rectal resection due to a benign condition, 9) rectal resection due to a recurrence of rectal cancer (previous anterior resection or another primary neoplasm), 10) rectal resection following a 'watch & wait' program, 11) emergency surgery, 12) previous derivative colostomy 13) inflammatory bowel disease.

DETAILED DESCRIPTION:
Accepting an alpha risk of 0.05 and a beta risk of 0.2 in a two-sided test, 45 subjects are necessary in first group and 45 in the second to recognize as statistically significant a difference greater than or equal to 2 units. The common standard deviation is assumed to be 3. It has been anticipated a drop-out rate of 20% Primary outcomes are LARS and Vaizey score. Secondary outcomes included are QLQ C30 and CR29, sexual function questionnaire (female/male), urinary function questionnaire and postoperative complications (Clavien-Dindo classification) Data will be collected in an online secure and protected repository (Castor edc). The planned study period is 2 years (September 2021 - September 2023).

It is essential to have a validated instrument that allows us to assess sphincter function and the different aspects of quality of life in operated patients, since increased survival in this pathology has led to greater importance in the evaluation functional outcome and quality of life; Furthermore, there are recent studies that speak of the direct relationship between these factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Informed consent
* Diagnosed with rectal cancer located below the peritoneal reflection, defined by preoperative MRI
* Open, laparoscopic, robotic or Transanal Total Mesorectal Excision (taTME) approaches
* Patients with/without derivative stoma
* Patients with/without neoadjuvant treatment

Exclusion Criteria:

* Upper rectal cancer, located above the peritoneal reflection
* Previous radical prostatectomy
* Previous pelvic radiotherapy
* Rectal resection without primary anastomosis
* Intraoperative findings of peritoneal carcinomatosis
* Stage IV disease
* Multivisceral or en-bloc resection, which includes uterus, prostate, vagina or bladder
* Rectal resection due to a benign condition
* Rectal resection due to a recurrence of rectal cancer (previous anterior resection or another primary neoplasm)
* Rectal resection following a 'watch & wait' program
* Emergency surgery
* Previous derivative colostomy
* Inflammatory bowel disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants that meet the criteria will be identified in each centre
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Low anterior resection syndrome (LARS) score | 2022
  LARS score from 0-42 where 0 means better outcomes
Vaizey score | 2022
  Incontinence score from 0-28 where 0 means better outcomes

SECONDARY OUTCOMES:
QLQ C30 | 2022
  Quality of Life questionnaire
QLQ CR29 | 2022
  Quality of life questionnaire, colorectal cancer related
Male sexual function | 2022
  IIEF questionnaire
Female sexual function | 2022
  FSFI questionnaires
Urinary function | 2022
  IPSS questionnaire
Postoperative complications | 2022
  Dindo-Clavien classification

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - University Clinic of Navarre, Madrid
  - University Hospital Gregorio Marañón, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bonjer HJ, Deijen CL, Abis GA, Cuesta MA, van der Pas MH, de Lange-de Klerk ES, Lacy AM, Bemelman WA, Andersson J, Angenete E, Rosenberg J, Fuerst A, Haglind E; COLOR II Study Group. A randomized trial of laparoscopic versus open surgery for rectal cancer. N Engl J Med. 2015 Apr 2;372(14):1324-32. doi: 10.1056/NEJMoa1414882. PMID 25830422
- [Result] Guillou PJ, Quirke P, Thorpe H, Walker J, Jayne DG, Smith AM, Heath RM, Brown JM; MRC CLASICC trial group. Short-term endpoints of conventional versus laparoscopic-assisted surgery in patients with colorectal cancer (MRC CLASICC trial): multicentre, randomised controlled trial. Lancet. 2005 May 14-20;365(9472):1718-26. doi: 10.1016/S0140-6736(05)66545-2. PMID 15894098
- [Result] 2017 European Society of Coloproctology (ESCP) collaborating group. An international multicentre prospective audit of elective rectal cancer surgery; operative approach versus outcome, including transanal total mesorectal excision (TaTME). Colorectal Dis. 2018 Sep;20 Suppl 6:33-46. doi: 10.1111/codi.14376. PMID 30255642
- [Result] Kim JY, Kim NK, Lee KY, Hur H, Min BS, Kim JH. A comparative study of voiding and sexual function after total mesorectal excision with autonomic nerve preservation for rectal cancer: laparoscopic versus robotic surgery. Ann Surg Oncol. 2012 Aug;19(8):2485-93. doi: 10.1245/s10434-012-2262-1. Epub 2012 Mar 21. PMID 22434245
- [Result] Park SY, Choi GS, Park JS, Kim HJ, Ryuk JP, Yun SH. Urinary and erectile function in men after total mesorectal excision by laparoscopic or robot-assisted methods for the treatment of rectal cancer: a case-matched comparison. World J Surg. 2014 Jul;38(7):1834-42. doi: 10.1007/s00268-013-2419-5. PMID 24366278
- [Result] Kim HJ, Choi GS, Park JS, Park SY, Yang CS, Lee HJ. The impact of robotic surgery on quality of life, urinary and sexual function following total mesorectal excision for rectal cancer: a propensity score-matched analysis with laparoscopic surgery. Colorectal Dis. 2018 May;20(5):O103-O113. doi: 10.1111/codi.14051. PMID 29460997
- [Result] Jayne D, Pigazzi A, Marshall H, Croft J, Corrigan N, Copeland J, Quirke P, West N, Rautio T, Thomassen N, Tilney H, Gudgeon M, Bianchi PP, Edlin R, Hulme C, Brown J. Effect of Robotic-Assisted vs Conventional Laparoscopic Surgery on Risk of Conversion to Open Laparotomy Among Patients Undergoing Resection for Rectal Cancer: The ROLARR Randomized Clinical Trial. JAMA. 2017 Oct 24;318(16):1569-1580. doi: 10.1001/jama.2017.7219. PMID 29067426
- [Result] Andolfi C, Umanskiy K. Appraisal and Current Considerations of Robotics in Colon and Rectal Surgery. J Laparoendosc Adv Surg Tech A. 2019 Feb;29(2):152-158. doi: 10.1089/lap.2018.0571. Epub 2018 Oct 16. PMID 30325690
- [Result] Sylla P, Rattner DW, Delgado S, Lacy AM. NOTES transanal rectal cancer resection using transanal endoscopic microsurgery and laparoscopic assistance. Surg Endosc. 2010 May;24(5):1205-10. doi: 10.1007/s00464-010-0965-6. Epub 2010 Feb 26. PMID 20186432
- [Result] Burch J, Taylor C, Wilson A, Norton C. Symptoms affecting quality of life after sphincter-saving rectal cancer surgery: A systematic review. Eur J Oncol Nurs. 2021 Jun;52:101934. doi: 10.1016/j.ejon.2021.101934. Epub 2021 Mar 22. PMID 33845303
- [Result] Christensen P, Im Baeten C, Espin-Basany E, Martellucci J, Nugent KP, Zerbib F, Pellino G, Rosen H; MANUEL Project Working Group. Management guidelines for low anterior resection syndrome - the MANUEL project. Colorectal Dis. 2021 Feb;23(2):461-475. doi: 10.1111/codi.15517. Epub 2021 Jan 24. PMID 33411977
- [Result] Li K, He X, Tong S, Zheng Y. Risk factors for sexual dysfunction after rectal cancer surgery in 948 consecutive patients: A prospective cohort study. Eur J Surg Oncol. 2021 Aug;47(8):2087-2092. doi: 10.1016/j.ejso.2021.03.251. Epub 2021 Mar 29. PMID 33832775
- [Derived] Tejedor P, Arredondo J, Pellino G, Pata F, Pastor C; PROCaRe study group. Patient Reported Outcomes following Cancer of the Rectum (PROCaRe): protocol of a prospective multicentre international study. Tech Coloproctol. 2023 Dec;27(12):1345-1350. doi: 10.1007/s10151-023-02865-4. Epub 2023 Sep 28. PMID 37770748